CLINICAL TRIAL: NCT03070509
Title: Pharmacokinetics of Lisdexamfetamine (Vyvanse®) in Post-bariatric Surgery Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Dakota State University (Other)
Collaborators: Shire (Industry); Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Responsible Party: Principal Investigator, Kristine Steffen, Associate Professor, North Dakota State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LIS-XXX
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Lisdexamfetamine
MeSH Terms: interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RYGB (Experimental): Single dose of lisdexamfetamine 50 mg in RYGB patients
  Interventions: Drug: Lisdexamfetamine
- Nonsurgical Controls (Experimental): Single dose of lisdexamfetamine 50 mg in non-surgical controls
  Interventions: Drug: Lisdexamfetamine

INTERVENTIONS:
Drug: Lisdexamfetamine — lisdexamfetamine 50 mg single dose

SUMMARY:
This study is being conducted to evaluate how the body absorbs and processes the medication lisdexamfetamine (Vyvanse®). Subjects who are 9-15 months post gastric bypass surgery will be invited to participate. Non-surgical controls will also be enrolled based on a matching criteria to post gastric bypass subjects. Participants will be asked to complete one 12-hour study day and complete one 24-hour post dosing blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects.
2. Between the ages of 18 and 60 years at the time of informed consent. *The upper age limit of 60 has been chosen as this medication carries some cardiovascular risk along with the fact that pharmacokinetics in elderly patients vary and may affect the homogeneity of the study.
3. Must be in good health as determined by physical exam, EKG, and medical history.

4a. Underwent RYGB 9-15 months prior (n=10 study completers) -or-

4b. Have not received bariatric surgery and are matched to the RYGB participants by BMI, age and sex (n= 10 study completers)

5. Women of child bearing potential must be practicing a medically acceptable method of birth control and have a negative pregnancy test at baseline.

6. No contraindications to receiving lisdexamfetamine in a single dose of 50 mg.

Exclusion Criteria:

1. Allergy to lisdexamfetamine or any of its constituents.
2. Candidates who are pregnant or nursing.
3. Candidates currently receiving a medication that interacts with lisdexamfetamine, including concurrent use of a stimulant.
4. Subjects who smoke or used any nicotine products in the last six months.
5. Subjects who have a positive urine drug screen for drugs of abuse.
6. Candidates that for any reason cannot comply with the requirements of the study procedures.
7. Candidates experiencing clinically significant or unstable neurological, hepatic, renal or cardiovascular disease on laboratory or baseline EKG screening or any medical disorder that would put the participant at increased risk in the judgement of the investigator or physician.
8. Candidates currently or with a past history of meeting diagnostic criteria for schizophrenia, schizoaffective disorder, bipolar disorder, or other psychotic illness.
9. Candidates with any history of drug abuse or dependence.
10. Candidates with any history of alcohol dependence, or current usage that puts the candidate at risk in the judgement of the investigator or study physician.
11. Candidates who have participated in an investigational drug study in the past 30 days.
12. Significant iron deficient anemia that may impact the pharmacokinetics of lisdexamfetamine.
13. Participant with a significantly and persistently elevated resting blood pressure (>140/90 mmHg) or pulse (>100 bpm) after repeated measurement.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Time Curve (AUC) of lisdexamfetamine | 24 hour collection
  The primary aim of this research is to provide a comparison of AUC associated with a single dose of lisdexamfetamine in Roux-en-Y Gastric Bypass and matched nonsurgical "control" subjects. Comparisons will be based upon lisdexamfetamine plasma concentrations obtained during the 24 hour sample collection window.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of lisdexamfetamine | 24 hour collection
  We will compare the Cmax of lisdexamfetamine associated with a single dose of lisdexamfetamine in Roux-en-Y Gastric Bypass and matched nonsurgical "control" subjects. Comparisons will be based upon lisdexamfetamine plasma concentrations obtained during the 24 hour sample collection window.
Time to Maximum Concentration (Tmax) of lisdexamfetamine | 24 hour collection
  We will compare the Tmax of lisdexamfetamine associated with a single dose of lisdexamfetamine in Roux-en-Y Gastric Bypass and matched nonsurgical "control" subjects. Comparisons will be based upon lisdexamfetamine plasma concentrations obtained during the 24 hour sample collection window.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuropsychiatric Research Institute, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No